CLINICAL TRIAL: NCT02424942
Title: A Two Part Protocol Using Double Blind Placebo Control to Assess the Safety, Tolerability, and Pharmacokinetics of Single Escalating Intra-articular Doses Followed by Assessment of Efficacy, Safety, Tolerability and Pharmacokinetics of a Single Intra-articular Dose of the TrkA Inhibitor, GZ389988, in Patients With Painful Osteoarthritis of the Knee
Brief Title: First-in-human Study With Ascending Single Intra-articular Doses of GZ389988 in Patients With Painful Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDU13828; 2014-004805-34 (EudraCT Number); U1111-1163-0806 (Other: UTN)
Record Dates: First submitted 2015-04-10; First posted 2015-04-23 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GZ389988 (Experimental): Single intraarticular injection of GZ389988 in the knee joint
  Interventions: Drug: GZ389988
- Placebo (Placebo Comparator): Single intraarticular injection of placebo for GZ389988 in the knee joint
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Pharmaceutical form:solvent for parenteral use
  Route of administration: intraarticular
  Arms: Placebo
Drug: GZ389988 — Pharmaceutical form:suspension for injection
  Route of administration: intraarticular
  Arms: GZ389988

SUMMARY:
Primary Objective:

To assess the safety and tolerability of ascending single intraarticular doses of GZ389988 in patients with painful osteoarthritis (OA) of the knee.

Secondary Objectives:

To assess the pharmacokinetic (PK) parameters of ascending single intraarticular doses of GZ389988 in patients with painful OA of the knee.

To obtain preliminary pharmacodynamic evaluation of ascending single intraarticular doses of GZ389988 in patients with painful OA of the knee.

DETAILED DESCRIPTION:
Screening will be performed within 28 days of dosing. Following the single dose of study medication, the study period for each patient will be 84 ± 7 days up to the end-of-study visit.

Total duration for one patient will be up to 17 weeks (up to the end-of-study visit), not including the long term observational safety follow-up by phone call for 12 additional weeks.

ELIGIBILITY:
Inclusion criteria :

* Men or women 40 to 60 years of age.
* Diagnosis of primary knee osteoarthritis, based upon the following:

  * Fulfilling the American College of Rheumatology Clinical and Radiographic criteria for OA (at least knee pain and osteophytes),
  * X-ray evidence within the last 6 months for Kellgren and Lawrence classification II to IV.
  * Western Ontario and McMaster Universities Arthritis Index (WOMAC) A1 Pain subscore (walking pain) between 50 and 90 using the 100-mm visual analog scale (VAS), corresponding to moderate to severe pain in the index knee, at both screening and baseline assessments at least 48 hours apart.
* Symptomatic for more than 6 months (if both symptomatic knees, at least for the most painful knee that will receive the study drug).
* Having given written informed consent prior to any procedure related to the study.
* Ambulatory with an active lifestyle and in good general health. (Assistive devices were allowed if used throughout a period of 3 months or more prior to screening, on the condition that they continued to be used throughout the study).
* A male who is sexually active must use a condom as part of a method of highly effective contraception (eg, condom + spermicide, and an additional contraceptive method used by the partner) during sexual intercourse with a women of childbearing potential for the duration of the study period up to the end-of-study visit and should not father a child in this period. Male patients also have to agree not to donate sperm for the duration of the study until the end-of-study visit.

Exclusion criteria:

* Women of childbearing potential.
* Pregnant or breastfeeding women.
* Any uncontrolled, chronic condition or laboratory finding which, in the opinion of the Investigator, could potentially put the patient at increased risk.
* Patients with clinically significant or uncontrolled hepatic, gastrointestinal, cardiovascular, respiratory, neurological (including diabetic neuropathy), psychiatric, hematological, renal, dermatological disease, or any other medical condition that might interfere with the evaluation of the investigational medicinal product (IMP) according to Investigator's medical judgment.
* Chondrocalcinosis.
* Fibromyalgia.
* Major depression.
* History or presence of drug or alcohol abuse (alcohol consumption >40 grams per day).
* Any patient who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Abnormal coagulation parameters: outside the range international normalized ratio (INR) 0.85-1.15, activated partial thromboplastin time >33 seconds, platelets <140 x 10^9/L.
* Moderate to severe renal impairment.
* Underlying hepatobiliary disease and/or alanine aminotransferase (ALT) >2 x upper limit of normal (ULN).
* High sensitivity C-reactive protein (hsCRP) >2 x ULN.
* Hemoglobin <10 g/dL, white blood cell count (WBC) <3 x 10^9/L.
* Positive result on any of the following tests: hepatitis B surface (HBsAg) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
* Secondary OA.
* Ipsilateral hip OA.
* Symptomatic contralateral knee OA with WOMAC A1 pain subscore (walking pain) >30 on 100-mm VAS.
* Prior history of osteonecrosis and/or rapidly progressive OA.
* Intraarticular injection within 3 months prior to inclusion.
* Unable to be maintained for at least 2 weeks prior to entry into study on paracetamol (No non-steroidal non-inflammatory drug [NSAID] use during the 12 weeks of the study; after the end-of-study visit [Day 84 ± 7] patients may be given an NSAID if necessary to provide better control of OA symptoms).
* Any IMP within 3 months prior to the study.
* Any knee MRI contraindication.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with adverse events | Up to Day 84 after single intraarticular dose of GZ389988
Proportion of patients with serious adverse events | 12 additional weeks after day 84 (by phone calls)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of GZ389988 single dose intraarticular (IA) | 24 timepoints up to Day 84
Area under the curve from time zero to last quantifiable concentration (AUClast) of single dose GZ389988 IA | 24 timepoints up to Day 84
Area under the curve (AUC) of single dose GZ389988 IA | 24 timepoints up to Day 84
Plasma elimination half-life (t1/2z) of single dose GZ389988 IA | 24 timepoints up to Day 84
Time to peak plasma concentration (tmax) of single dose GZ389988 IA | 24 timepoints up to Day 84
Time curve from administration to last measurement (tlast) of single dose GZ389988 IA | 24 timepoints up to Day 84
Apparent volume of distribution (Vz/F) of single dose GZ389988 IA | 24 timepoints up to Day 84
Apparent total body clearance(CL/F) of single dose GZ389998 IA | 24 timepoints up to Day 84
Synovial fluid concentrations (if possible) of single dose GZ389988 IA | 3 timepoints up to Day 84
Change from baseline in WOMAC index (total score) | Over 1, 2, 3, 4, 6, 8, 10, and 12 weeks following the single intraarticular injection
Change from baseline in WOMAC pain (including WOMAC A1 pain subscores) | Over 1, 2, 3, 4, 6, 8, 10, and 12 weeks following the single intraarticular injection
Change from baseline in WOMAC stiffness subscore | Over 1, 2, 3, 4, 6, 8, 10, and 12 weeks following the single intraarticular injection
Change from baseline in WOMAC physical function subscore | Over 1, 2, 3, 4, 6, 8, 10, and 12 weeks following the single intraarticular injection

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 276001, Berlin, Germany